CLINICAL TRIAL: NCT06621888
Title: Investigating The Effects Of Full-Spectrum Medicinal Cannabis Plant Extract 0.08% THC (NTI164) On Paediatric Acute-onset Neuropsychiatric Syndrome (PANS)
Acronym: CannaPANS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTIPANS1; ACTRN12622001419752 (Other: ANZCTR)
Record Dates: First submitted 2024-09-11; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: PANS Pediatric Acute-Onset Neuropsychiatric Syndrome
MeSH Terms: conditions — Pediatric acute-onset neuropsychiatric syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active NTI164 Group (Experimental): Participants in this group receive Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164) to treat pediatric acute-onset neuropsychiatric syndrome (PANS). The treatment begins with an up-titration phase where doses start at 5 mg/kg daily and increase to a maximum of 20 mg/kg. This is followed by an 8-week treatment phase at the maximum tolerated dose. Participants have the option to extend this phase up to 54 weeks. The study concludes with a down-titration phase, gradually reducing the dose over 4 weeks. Efficacy is assessed through psychological questionnaires and immune function tests.
  Interventions: Drug: NTI164

INTERVENTIONS:
Drug: NTI164 — This intervention uses Full-Spectrum Medicinal Cannabis Plant Extract with a low THC concentration of 0.08% (NTI164), specifically formulated to treat pediatric acute-onset neuropsychiatric syndrome (PANS). The dosing regimen is carefully structured to increase from an initial 5 mg/kg per day up to a maximum of 20 mg/kg, tailored to individual tolerance levels. This gradual titration and the option to extend treatment up to 54 weeks distinguishes it from other interventions that may use different concentrations of THC or shorter treatment durations. The efficacy of NTI164 is rigorously assessed through psychological evaluations and biomarker analyses.

SUMMARY:
This study investigates the effectiveness of a medicinal cannabis extract (NTI164) with 0.08% THC in treating children with pediatric acute-onset neuropsychiatric syndrome (PANS) over a period of 18 to 54 weeks. Participants, aged 18 to 54, will start with a daily dose of 5mg/kg, gradually increasing to a maximum of 20mg/kg over four weeks. After reaching their maximum tolerated dose, they will maintain this dose for eight weeks, with an option to extend up to 54 weeks. The study will measure the treatment's efficacy using questionnaires on emotional and behavioral changes, and verify the results with whole blood RNA sequencing to assess immune dysfunction.

DETAILED DESCRIPTION:
This open-label study spans 18 to 54 weeks and aims to assess the efficacy of Full-Spectrum Medicinal Cannabis Plant Extract containing 0.08% THC (NTI164) for treating pediatric acute-onset neuropsychiatric syndrome (PANS) in children. The main objective is to evaluate how effective the NTI164 treatment is over the specified duration.

The study protocol involves several phases:

1. **Up-titration phase:** Participants will start with a daily dosage of 5 mg/kg of NTI164, incrementally increasing this dose over a four-week period until reaching either the maximum tolerated dose or 20 mg/kg per day.
2. **Treatment phase:** Following the up-titration, participants will continue at their maximum tolerated dose for eight weeks.
3. **Extension phase:** After the initial eight-week treatment phase, participants have the option to continue at their maximum dose for up to an additional 46 weeks, totaling a possible 54 weeks of treatment.
4. **Down-titration phase:** At the conclusion of the treatment or extension phases, the dosage will be gradually reduced by 5 mg/kg over four weeks until the participant's involvement in the study ends.

The effectiveness of NTI164 will be monitored through both participant- and psychologist-led questionnaires, which are designed to track changes in the emotions and behavior of the patients with PANS. Additionally, the study will employ whole blood RNA sequencing as a method to validate the presence of an immune dysfunction signature, aiming to provide a biomarker for response to treatment. This comprehensive approach seeks to ensure a thorough evaluation of NTI164's potential benefits in alleviating the symptoms of PANS.

ELIGIBILITY:
Inclusion Criteria:

* 1 - 17 years of age
* Patients who fulfil PANS criteria
* Acute onset of OCD or severely restricted food intake
* Concurrent presentation of additional neuropsychiatric symptoms from at least 2 of the following 7 categories: anxiety, emotional lability/depression, irritability, aggression or severely oppositional behaviours, behavioural regression, deterioration in school performance, sensory or motor abnormalities (e.g. tics), somatic symptoms (e.g. sleep disturbances, enuresis or increase in urinary frequency)
* Symptoms not better explained by a known neurologic or medical disorder (e.g. Sydenham's chorea)
* RCADS-P scores of >65 (a scale of anxiety, social phobia, panic disorder, OCD, and low mood, a score of >65 infers moderate-significant impairment)
* Other patient medications (e.g. anti-psychotics) must be stable for at least 12 weeks prior to trial participation

Exclusion Criteria:

* Infection and/or antibiotic use in the 2 weeks prior to trial participation (i.e. baseline blood tests and commencement of NTI164)
* Recent changes to other patient medication (e.g. addition or escalation of anxiolytics, anti-depressants etc; medication dosage must be stable for at least 12 weeks prior to trial participation)
* Intellectual disability preventing adequate assent from patient, or that would affect reporting throughout trial; patients with intellectual disability must still have the capacity to verbalise their symptoms/experiences
* Ongoing immunomodulating or immunosuppressive treatment use in the previous 12 weeks, including steroids, IVIG, antibiotics, low-dose naltrexone, mycophenolate, Rituximab etc.
* Currently using or has used recreational or medicinal cannabis or cannabinoid-based medications (e.g. Sativex ®, Epidiolex ®) in the previous 12 weeks and/or is unwilling or unable to abstain for the duration of the trial
* Underlying renal impairment, cardiovascular issues (e.g. arrhythmia), current or previous thrombosis
* Impaired hepatic function, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN) or total bilirubin (TBL) > 2 x ULN; this criterion can only be confirmed once baseline laboratory results are available and participants who fail this criterion will not proceed in this study
* Other diagnosed neurological condition likely to be contributing to OCD/neuropsychiatric symptoms (e.g. Huntington's disease)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale-Improvement | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The CGI-I (Clinical Global Impressions - Improvement) scale rates patient improvement on a scale from 1 to 7. Lower scores indicate better improvement.
Revised Childrens Anxiety and Depression Scale-Parent Version | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The RCADS-P (Revised Child Anxiety and Depression Scale - Parent Version) assesses anxiety and depression in children, with individual item scores ranging from 0 to 3. Higher scores indicate more severe symptoms, meaning lower scores suggest better emotional well-being.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The Yale Global Tic Severity Scale (YGTSS) measures the severity of tics in individuals, with individual item scores ranging from 0 to 5 for both motor and vocal tics. Higher scores indicate more severe tics and lower scores reflect better tic control.
Children's Yale-Brown Obsessive-Compulsive Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) assesses the severity of obsessive-compulsive symptoms in children, with individual item scores ranging from 0 to 4. Higher scores indicate more severe symptoms and lower scores suggest better symptom control.
Conners Scale | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The Conners' Scale measures behavioural problems, with individual item scores ranging from 0 to 3. Higher scores indicate more severe behavioural issues and lower scores reflect better behavioural functioning.
EQ-5D-Y | Baseline (pre-dose), 4, 12, 16 weeks post-commencement of treatment. Additional timepoints for Extension phase: Weeks 28, 40, 52 post-commencement of treatment.
  The EQ-5D-Y (EuroQol Five-Dimension Youth) is a measure of health-related quality of life in children and adolescents. It assesses five dimensions, with individual item scores ranging from 1 to 3. A higher score indicates more health-related difficulties, meaning lower scores reflect better quality of life.
Blood Transcriptomic Signature | Baseline (pre-dose) and 16 weeks post-commencement of treatment.
  The Blood Transcriptomic Signature outcome assesses changes in gene expression in PANS children post-NTI164 treatment, compared to baseline and controls. RNA sequencing of blood samples will identify modifications in the transcriptomic profile, providing insights into the treatment's impact on molecular processes.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - The Childrens Hospital at Westmead, Sydney, New South Wales
  - Monash Children's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as per commercial in confidence restrictions.